CLINICAL TRIAL: NCT03490032
Title: A Phase 1/2 Open-label, Multi-center, Safety and Tolerability Study of a Single Dose of 68Ga-PSMA-R2 in Patients With Biochemical Relapse (BR) and Metastatic Prostate Cancer (mPCa)
Brief Title: 68Ga-PSMA-R2 in Patients With Biochemical Relapse (BR) and Metastatic Prostate Cancer (mPCa)
Acronym: PROfind
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: A206D-A01-001; CAAA502A12101 (Other: Novartis)
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostatic Neoplasms; Cancer of Prostate; Cancer of the Prostate; Neoplasms, Prostate; Prostate Cancer; Prostatic Cancer; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Diseases; PSMA; Prostate-specific membrane antigen; Gallium radioisotope 68; 68Ga-PSMA-R2; 68Ga-PSMA ligand
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Diseases

STUDY DESIGN:
Intervention Model Description: Phase I: characterize PK and dosimetry Phase II: diagnostic potential in 2 groups
  1. Prostate Cancer in biochemical relapse, and
  2. Metastatic Prostate Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) (Experimental): All eligible participants received recommended dose of [68Ga]-PSMA-R2 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
  Interventions: Drug: [68Ga]-PSMA-R2
- Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) (Experimental): All eligible participants received recommended dose of [68Ga]-PSMA-R2 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
  Interventions: Drug: [68Ga]-PSMA-R2
- Metastatic Prostate Cancer (mPCa) (Phase II) (Experimental): All eligible participants received recommended dose of [68Ga]-PSMA-R2 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
  Interventions: Drug: [68Ga]-PSMA-R2

INTERVENTIONS:
Drug: [68Ga]-PSMA-R2 — radio-labelled PSMA ligand

SUMMARY:
This was an open-label, multicenter, single dose, Phase I/II study to evaluate the safety and tolerability of a single administration of 3 mega Becquerel (MBq)/kg, but not less than 150 MBq and not more than 250 MBq, of 68^Ga-PSMA-R2 in adult male patients with biochemical relapse (BR) and metastatic prostate cancer (mPCa).

DETAILED DESCRIPTION:
This study consisted of 2 parts.

* During the first part (Phase I) of the study, 6 subjects with biochemically recurrent prostate cancer (PCa) received the investigational product (IP) and remained at the site for approximately 6 hours post-administration in order to assess the PK, biodistribution versus time, and dosimetry for critical organs. Subjects received a single dose of 3 MBq/kg, (>=150 and =<250 MBq), of 68^Ga-PSMA-R2 intravenously. Serial blood and urine samples were collected for PK characterization and dosimetry and whole-body PET/CT were acquired at selected time points (0 to 4 hours) to determine organ and tumor absorbed doses. Safety assessments were conducted after IP administration on Day 1, and during follow-up on Days 7 and 28.
* In the second part of the study (Phase II), 2 groups of 12 subjects were enrolled (subjects with PCa in biochemical recurrence [PCa-BR], and subjects with prostate cancer in the metastatic stage [mPCa]). Based on the preliminary data analysis from the Phase I part of the study provided sufficient dosimetry data, all subjects underwent the whole body PET/CT imaging optimized for time (up to 2 time points) according to the data analysis from the Phase I part of the study.

This study was comprised of 4 clinical visits and conducted in 3 study periods: screening, administration/imaging, and safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Males 18 years or older.
2. Signed and dated written informed consent by the subject prior to any study-specific procedures.
3. Histologically confirmed adenocarcinoma of the prostate, defined as follows:

   1. Biochemical recurrence: defined as PSA is ≥0.2 ng/mL after radical prostatectomy or PSA nadir plus 2 ng/mL after radiation therapy with corresponding CT/MRI or bone scan revealing absence of local recurrence or metastatic lesions.

      OR
   2. Metastatic disease: defined as both, castration-sensitive or castration-resistant mPCa (presence of at least 1 metastatic lymph node, visceral metastasis and/or bone metastasis).
   3. At least 2 weeks must have elapsed between last anticancer treatment administration and the administration of the imaging product, 68Ga-PSMA-R2.
4. Prior major surgery must be at least 12 weeks prior to study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2, with a life expectancy ≥6 months.
6. Adequate bone marrow reserve and organ function as demonstrated by complete blood count, and biochemistry in blood and urine at Screening:

   1. Hemoglobin (Hb): >8 g/dL
   2. Platelet count of >50.000/mm3
7. Serum creatinine <1.5*upper limit normal (ULN) or estimated glomerular filtration rate (eGFR) >50 mL/min based upon The Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
8. For male subjects with partners of childbearing potential, agreement to use barrier contraceptive method (condom) and to continue its use for 28 days after IP administration.

Exclusion Criteria:

1. Pathological finding consistent with small cell, neuroendocrine carcinoma of the prostate or any other histologies different than adenocarcinoma.
2. Administered a radioisotope =<10 physical half-lives prior to the day of PET/CT.
3. Current severe urinary incontinence, hydronephrosis, severe voiding dysfunction, or need of indwelling/condom catheters.
4. Uncontrolled pain or incompatibility that results in subject's lack of compliance with imaging procedures.
5. Other known coexisting malignancies except non-melanoma skin or low grade superficial bladder cancer unless definitively treated and proven no evidence of recurrence for 5 years.
6. Subject with known incompatibility to CT scans.
7. Any evidence of severe or uncontrolled systemic or psychiatric diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol, or active infection including human immunodeficiency virus (HIV) and untreated hepatitis B, hepatitis C. Screening for chronic conditions was not required.
8. Subjects who have received any investigational agent within the last 28 days were excluded from participation in this study.
9. Any acute toxicity due to prior chemotherapy and/or radiotherapy that has not resolved according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Studies.
10. Known allergy, hypersensitivity, or intolerance to the IP or its excipients.
11. Subject unlikely to comply with study procedures, restrictions and requirements and judged by the investigator to be unsuitable for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Pheonix Molecular Imaging Center, Phoenix, Arizona
  - University of California, San Francisco (UCSF), San Francisco, California
  - Smilow Cancer Center at Yale New Haven, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
  - National Institutes of Health, Warren Grant Magnusen Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in the USA (Phase I: 1 site; Phase II: 4 sites)
Period: Overall Study
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Started (All enrolled patients were included in the Full Analysis Set (FAS)) | 6 | 12 | 12
Completed | 5 | 12 | 12
Not Completed | 1 | 0 | 0
Not completed — family issue (child custody) | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II) | Total
Number analyzed (Participants) | 6 | 12 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (7.91) | 69.1 (6.53) | 68.6 (10.00) | 68.3 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 12 | 12 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 1 | 0 | 1
  White | 6 | 10 | 11 | 27
  Other | 0 | 1 | 1 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classifies participants according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). ECOG PS: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Grade 0 | 6 | 9 | 6 | 21
    > = Grade 1 | 0 | 3 | 6 | 9
Prostate-specific antigen (PSA) levels [Mean (Standard Deviation); unit: ng/mL] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  ng/mL | 1.68 (1.329) | 3.72 (6.461) | 38.56 (66.603) | 17.25 (44.861)
Time since first prostate cancer diagnosis [Mean (Standard Deviation); unit: Months] — Time since first prostate cancer diagnosis is defined as (date of screening - date of first prostate cancer diagnosis + 1) / 30.4375.
  Months | 79.2 (46.44) | 86.8 (78.07) | 96.1 (84.80) | 88.8 (73.41)
Time since first metastasis [Mean (Standard Deviation); unit: Months] — Time since first metastasis is defined as (date of screening - date of first metastasis + 1)/ 30.4375.
  Months | 79.2 (46.44) | 86.8 (78.07) | 96.1 (84.80) | 88.8 (73.41)
Time since disease progression [Mean (Standard Deviation); unit: Months] — Time since disease progression is defined as (date of screening - date of disease progression + 1)/ 30.4375.
  Months | 34.7 (33.02) | 1.2 (1.55) | 0.8 (0.65) | 5.8 (16.01)
Number of patients by castration type [Count of Participants; unit: Participants]
  Surgery | 0 | 10 | 4 | 14
  Pharmacological | 1 | 3 | 11 | 15
  Not Applicable | 1 | 1 | 0 | 2
Number of patients by Primary and Secondary Gleason score [Count of Participants; unit: Participants] — The Gleason score is based on biopsy samples taken from the prostate. Both a primary and a secondary pattern of tissue organization are identified. The primary pattern represents the most common tissue pattern seen in the tumor, and the secondary pattern represents the next most common pattern. Each pattern is given a grade from 1 to 5, with 1 looking the most like normal prostate tissue and 5 looking the most abnormal. The two grades are then added to give a Gleason score.
  Participants
    Primary Gleason score=3 &Secondary Gleason score=3 | 0 | 2 | 2 | 4
    Primary Gleason score=3 &Secondary Gleason score=4 | 2 | 4 | 0 | 6
    Primary Gleason score=4 &Secondary Gleason score=3 | 2 | 4 | 3 | 9
    Primary Gleason score=4 &Secondary Gleason score=4 | 0 | 1 | 3 | 4
    Primary Gleason score=4 &Secondary Gleason score=5 | 2 | 1 | 4 | 7
Number of patients by Total Gleason score (>=6) [Count of Participants; unit: Participants] — Gleason score can range from 2-10. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly. Scores of 6 (or less) describe cancer cells that look similar to normal cells and suggest that the cancer is likely to grow slowly. A score of 7 suggests an intermediate risk for aggressive cancer. Scores of 8 (or higher) describe cancers that are likely to spread more rapidly, these cancers are often referred to as poorly differentiated or high grade.
  Participants
    6 | 0 | 2 | 2 | 4
    7 | 4 | 8 | 3 | 15
    8 | 0 | 1 | 3 | 4
    9 | 2 | 1 | 4 | 7
    10 | 0 | 0 | 0 | 0
Baseline Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  kilogram (kg) | 91.48 (18.091) | 87.03 (18.838) | 93.20 (11.402) | 90.29 (15.890)
Baseline Height [Mean (Standard Deviation); unit: centimeter (cm)] — Baseline is defined as the last measurement prior to Investigational Medicinal Product (IMP) administration.
  centimeter (cm) | 183.00 (5.030) | 177.96 (6.596) | 177.03 (5.927) | 178.65 (6.281)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were collected from first dosing (single administration, Day 1) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent. The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: dosing through 28 days post-dose
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Participants
  Treatment-Emergent Adverse Events (TEAEs) | 1 | 4 | 2
  Serious TEAEs | 0 | 1 | 0
  Deaths Due to AEs | 0 | 0 | 0

2. Secondary Outcome: Phase I: Decay Corrected Tissue Time-activity Curves (TACs) From 68Ga-PSMA-R2 PET/CT Images in Normal Organs
Description: PET/CT scans were performed at approximately 20 to 30 min and at 1, 2, 3 to 4 hours postinjection. Time activity curves (TACs) for various organs (Brain, Heart Wall, Kidney, Lacrimal Gland, Liver, Lungs, Salivary Gland, Spleen and Thyroid) were produced as decay-corrected tissue of injected activity (mSv/MBq) per organ. Only descriptive analysis performed.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (20-30 min post-injection, 1 hour, 2 hours and 3-4 hours post-injection)
Population: Full Analysis Set (FAS). Only participants with a value at each post-injection timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mSv/MBq
  Brain@20-30 minutes post-injection | 0.002196 (0.0009359)
  Brain@1 hour post-injection | 0.001913 (0.0003011)
  Brain@2 hours post-injection | 0.001310 (0.0005902)
  Brain@3-4 hours post-injection | 0.001279 (0.0007786)
  Heart Wall@20-30 minutes post-injection | 0.009010 (0.0014472)
  Heart Wall@1 hour post-injection | 0.006371 (0.0012260)
  Heart Wall@2 hours post-injection | 0.004330 (0.0014781)
  Heart Wall@3-4 hours post-injection | 0.003209 (0.0014961)
  Kidney@20-30 minutes post-injection | 0.033219 (0.0140235)
  Kidney@1 hour post-injection | 0.022069 (0.0090106)
  Kidney@2 hours post-injection | 0.018424 (0.0068331)
  Kidney@3-4 hours post-injection | 0.015772 (0.0069341)
  Lacrimal Gland@20-30 minutes post-injection | 0.000016 (0.0000023)
  Lacrimal Gland@1 hour post-injection | 0.000016 (0.0000051)
  Lacrimal Gland@2 hours post-injection | 0.000015 (0.0000045)
  Lacrimal Gland@3-4 hours post-injection | 0.000014 (0.0000074)
  Liver@20-30 minutes post-injection | 0.040546 (0.0098781)
  Liver@1 hour post-injection | 0.030958 (0.0073605)
  Liver@2 hours post-injection | 0.023145 (0.0083627)
  Liver@3-4 hours post-injection | 0.018128 (0.0081345)
  Lungs@20-30 minutes post-injection | 0.010066 (0.0017280)
  Lungs@1 hour post-injection | 0.007535 (0.0013048)
  Lungs@2 hours post-injection | 0.005023 (0.0015987)
  Lungs@3-4 hours post-injection | 0.003601 (0.0016623)
  Salivary Gland@20-30 minutes post-injection | 0.002001 (0.0004118)
  Salivary Gland@1 hour post-injection | 0.001585 (0.0004877)
  Salivary Gland@2 hours post-injection | 0.001282 (0.0006661)
  Salivary Gland@3-4 hours post-injection | 0.001032 (0.0005455)
  Spleen@20-30 minutes post-injection | 0.003712 (0.0010597)
  Spleen@1 hour post-injection | 0.002645 (0.0008966)
  Spleen@2 hours post-injection | 0.001724 (0.0007601)
  Spleen@3-4 hours post-injection | 0.001264 (0.0006056)
  Thyroid@20-30 minutes post-injection: number analyzed (Participants) | 1
  Thyroid@20-30 minutes post-injection | 0.000378 (NA) — Only one participant analyzed
  Thyroid@1 hour post-injection: number analyzed (Participants) | 1
  Thyroid@1 hour post-injection | 0.000266 (NA) — Only one participant analyzed
  Thyroid@2 hours post-injection: number analyzed (Participants) | 1
  Thyroid@2 hours post-injection | 0.000201 (NA) — Only one participant analyzed
  Thyroid@3-4 hours post-injection: number analyzed (Participants) | 1
  Thyroid@3-4 hours post-injection | 0.000128 (NA) — Only one participant analyzed

3. Secondary Outcome: Phase I: Urinary Excretion of [68Ga]-PSMA-R2
Description: Urine samples were collected (up to 6 hours after dosing) for activity-based pharmacokinetics characterization. The apparent systemic clearance for the analyte in urine (Cl) was summarized with descriptive statistics.
Time Frame: 0 to 6 hours post-dose
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mL/hr | 5870 (1820)

4. Secondary Outcome: Phase I: Half-life of 68Ga-PSMA-R2 in Blood
Description: Serial blood samples were collected (up to 6 hours after dosing) for activity-based pharmacokinetics characterization. The half-life (T^1/2) for the analyte in blood was summarized with descriptive statistics.
Time Frame: 0 to 6 hours post-dose
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
Hour | 2.83 (0.868)

5. Secondary Outcome: Phase I: Non-decay Corrected Tissue Time-activity Curves (TACs) From 68Ga-PSMA-R2 PET/CT Images in Normal Organs
Description: PET/CT scans were performed at approximately 20 to 30 min and at 1, 2, 3 to 4 hours postinjection. Time activity curves (TACs) for the various organs were produced as non-decay-corrected fraction of injected activity (mSv/MBq) per organ. Only descriptive analysis performed.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (20-30 min post-injection, 1 hour, 2 hours and 3-4 hours post-injection)
Population: Full Analysis Set (FAS). Only participants with a value at each post-injection timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mSv/MBq
  Brain@20-30 minutes post-injection | 0.001686 (0.0007242)
  Brain@1 hour post-injection | 0.001046 (0.0000814)
  Brain@2 hours post-injection | 0.000423 (0.0001630)
  Brain@3-4 hours post-injection | 0.000222 (0.0000924)
  Heart Wall@20-30 minutes post-injection | 0.006914 (0.0011156)
  Heart Wall@1 hour post-injection | 0.003484 (0.0004766)
  Heart Wall@2 hours post-injection | 0.001332 (0.0002056)
  Heart Wall@3-4 hours post-injection | 0.000542 (0.0001255)
  Kidney@20-30 minutes post-injection | 0.025506 (0.0107777)
  Kidney@1 hour post-injection | 0.012059 (0.0043426)
  Kidney@2 hours post-injection | 0.005825 (0.0015596)
  Kidney@3-4 hours post-injection | 0.002766 (0.0006581)
  Lacrimal Gland@20-30 minutes post-injection | 0.000012 (0.0000019)
  Lacrimal Gland@1 hour post-injection | 0.000009 (0.0000022)
  Lacrimal Gland@2 hours post-injection | 0.000005 (0.0000011)
  Lacrimal Gland@3-4 hours post-injection | 0.000002 (0.0000008)
  Liver@20-30 minutes post-injection | 0.031128 (0.0076342)
  Liver@1 hour post-injection | 0.016949 (0.0032692)
  Liver@2 hours post-injection | 0.007172 (0.0014994)
  Liver@3-4 hours post-injection | 0.003087 (0.0006828)
  Lungs@20-30 minutes post-injection | 0.007729 (0.0013599)
  Lungs@1 hour post-injection | 0.004149 (0.0006660)
  Lungs@2 hours post-injection | 0.001573 (0.0002652)
  Lungs@3-4 hours post-injection | 0.000631 (0.0001601)
  Salivary Gland@20-30 minutes post-injection | 0.001536 (0.0003192)
  Salivary Gland@1 hour post-injection | 0.000859 (0.0002093)
  Salivary Gland@2 hours post-injection | 0.000386 (0.0001469)
  Salivary Gland@3-4 hours post-injection | 0.000173 (0.0000550)
  Spleen@20-30 minutes post-injection | 0.002849 (0.0008140)
  Spleen@1 hour post-injection | 0.001444 (0.0004213)
  Spleen@2 hours post-injection | 0.000536 (0.0001640)
  Spleen@3-4 hours post-injection | 0.000217 (0.0000567)
  Thyroid@20-30 minutes post-injection: number analyzed (Participants) | 1
  Thyroid@20-30 minutes post-injection | 0.000289 (NA) — Only one participant analyzed
  Thyroid@1 hour post-injection: number analyzed (Participants) | 1
  Thyroid@1 hour post-injection | 0.000136 (NA) — Only one participant analyzed
  Thyroid@2 hours post-injection: number analyzed (Participants) | 1
  Thyroid@2 hours post-injection | 0.000057 (NA) — Only one participant analyzed
  Thyroid@3-4 hours post-injection: number analyzed (Participants) | 1
  Thyroid@3-4 hours post-injection | 0.000020 (NA) — Only one participant analyzed

6. Secondary Outcome: Phase I: Residence Times in Normal Organs
Description: Residence times of radiation in normal organs were summarized with descriptive statistics.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS). For each parameter, only participants with a value are included in the analysis.
Measure: Mean (Standard Deviation); unit: MBq-hr/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
MBq-hr/MBq
  Brain | 0.002895 (0.0009849)
  Heart | 0.010459 (0.0014152)
  Kidney | 0.039360 (0.0133500)
  Lacrimal Gland | 0.000027 (0.0000052)
  Liver | 0.050735 (0.0103951)
  Lungs | 0.012084 (0.0019321)
  Salivary Gland | 0.002594 (0.0006622)
  Spleen | 0.004291 (0.0012416)
  Thyroid: number analyzed (Participants) | 1
  Thyroid | 0.000424 (NA) — Only one participant analyzed
  Urinary Bladder | 0.092947 (0.0453608)
  Remainder | 1.417135 (0.0582923)

7. Secondary Outcome: Phase I: Absorbed Dose of 68Ga-PSMA-R2
Description: Absorbed radiation dose of 68Ga-PSMA-R2 in target organs were summarized with descriptive statistics.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: mGy/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mGy/MBq
  Brain | 0.002563 (0.000336)
  Heart | 0.018417 (0.0020094)
  Kidney | 0.060683 (0.0190588)
  Lacrimal Gland | 0.008065 (0.0015741)
  Liver | 0.017417 (0.0029976)
  Lungs | 0.007967 (0.0007718)
  Red Marrow | 0.010700 (0.0002280)
  Salivary Gland | 0.015600 (0.0032012)
  Spleen | 0.017333 (0.0037109)
  Urinary Bladder | 0.120317 (0.0517023)

8. Secondary Outcome: Phase I: Whole-body Dose of 68Ga-PSMA-R2
Description: The whole-body dose of 68Ga-PSMA-R2 was summarized with descriptive statistics.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: mGy/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mGy/MBq | 0.013800 (0.0000632)

9. Secondary Outcome: Phase I: Effective Dose of 68Ga-PSMA-R2
Description: The effective dose of 68Ga-PSMA-R2 was summarized with descriptive statistics.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I)
Number analyzed (Participants) | 6
mSv/MBq | 0.014583 (0.0019343)

10. Secondary Outcome: Standard Uptake Value (SUV) Mean and Max in Lesions Detected by PET Scans by Timepoint
Description: Targeting properties of 68Ga-PSMA-R2 were evaluated by semi-quantitatively assessing radiotracer uptake at lesion level, identified via PET/CT imaging (4 scans). The SUVmean and SUVmax (g/mL) of each lesion were calculated and reported by lesion location with summary statistics at all imaging time points.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Standard Uptake Value (SUV)
  PET (1hr): SUVmax (lesion) | 4.493 (1.4060) | 4.421 (1.4512) | 6.725 (5.5327)
  PET (1hr): SUVmean (background) | 0.980 (0.0283) | 0.643 (0.2318) | 0.750 (0.3002)
  PET (2hr): SUVmax (lesion) | 3.767 (1.1493) | 5.098 (1.8597) | 6.846 (4.7745)
  PET (2hr): SUVmean (background) | 0.630 (0.3145) | 0.651 (0.2817) | 0.550 (0.1948)

11. Secondary Outcome: Tumor to Background Ratio (TBR) of Lesions Detected by PET Scans by Timepoint
Description: Targeting properties of 68Ga-PSMA-R2 were evaluated by semi-quantitatively assessing radiotracer uptake at lesion level, identified via PET/CT imaging (4 scans). The lesion Tumor to Background Ratio (TBR) was defined as SUVmax(lesion) / SUVmean(gluteal or thigh) was calculated and reported by lesion location with summary statistics at all imaging time points.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Ratio
  PET (1hr): TBR | 4.520 (1.3558) | 7.464 (3.0364) | 11.141 (10.6283)
  PET (2hr): TBR | 5.694 (1.7104) | 7.780 (3.6034) | 12.588 (9.1146)

12. Secondary Outcome: Standard Uptake Value (SUV) Mean and Max in Lesions Detected by PET Scans and Also Detected by Conventional Scans by Timepoint
Description: as for outcome 10
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS). Only participants with at least 1 positive lesion detected by conventional scan and at least 1 positive lesion detected by PET included in the analysis.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Standard Uptake Value (SUV)
  PET (1hr): SUVmax (lesion): number analyzed (Participants) | 0 | 0 | 12
  PET (1hr): SUVmax (lesion) |  |  | 7.087 (4.9133)
  PET (1hr): SUVmean (background): number analyzed (Participants) | 0 | 0 | 12
  PET (1hr): SUVmean (background) |  |  | 0.689 (0.1955)
  PET (2hr): SUVmax (lesion): number analyzed (Participants) | 0 | 0 | 12
  PET (2hr): SUVmax (lesion) |  |  | 7.647 (5.3409)
  PET (2hr): SUVmean (background): number analyzed (Participants) | 0 | 0 | 12
  PET (2hr): SUVmean (background) |  |  | 0.541 (0.2234)

13. Secondary Outcome: Tumor to Background Ratio (TBR) of Lesions Detected by PET Scans and Also Detected by Conventional Scans by Timepoint
Description: as for outcome 11
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Ratio
  PET (1hr): TBR: number analyzed (Participants) | 0 | 0 | 12
  PET (1hr): TBR |  |  | 11.573 (10.2632)
  PET (2hr): TBR: number analyzed (Participants) | 0 | 0 | 12
  PET (2hr): TBR |  |  | 14.880 (10.1991)

14. Secondary Outcome: Standard Uptake Value (SUV) Mean and Max in Lesions Detected by PET Scans and Not Detected by Conventional Scans by Timepoint
Description: as for outcome 10
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Standard Uptake Value (SUV)
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Standard Uptake Value (SUV)
  PET (1hr): SUVmax (lesion) | 4.493 (1.4060) | 4.421 (1.4512) | 6.578 (5.8224)
  PET (1hr): SUVmean (background) | 0.980 (0.0283) | 0.643 (0.2318) | 0.723 (0.3020)
  PET (2hr): SUVmax (lesion) | 3.767 (1.1493) | 5.098 (1.8597) | 6.566 (4.5956)
  PET (2hr): SUVmean (background) | 0.630 (0.3145) | 0.651 (0.2817) | 0.581 (0.2119)

15. Secondary Outcome: Tumor to Background Ratio (TBR) of Lesions Detected by PET Scans and Not Detected by Conventional Scans by Timepoint
Description: as for outcome 11
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Ratio
  PET (1hr): TBR | 4.520 (1.3558) | 7.464 (3.0364) | 10.965 (10.9067)
  PET (2hr): TBR | 5.694 (1.7104) | 7.780 (3.6034) | 11.788 (8.6914)

16. Secondary Outcome: Patient Level Agreement of 68Ga-PSMA-R2 PET Imaging Relative to Conventional Techniques in Prostate Cancer Patients
Description: The subject-level positive percent agreement, negative percent agreement, and overall percent agreement was calculated based on the number of subjects with at least 1 positive lesion detected by conventional scan or at least 1 positive lesion detected by PET scan. These percent agreements were calculated as follows:
  * Positive percent agreement: a/(a+c) × 100
  * Negative percent agreement: d/(b+d) × 100
  * Overall percent agreement: (a+d)/(a+b+c+d) × 100
  Where:
  * a = number of subjects with at least 1 positive lesion detected by conventional scan and at least 1 positive lesion detected by PET scan
  * b = number of subjects with at least 1 positive lesion detected by PET scan that was not correlated with conventional scan
  * c = number of subjects with at least 1 positive lesion detected by conventional scan that was not correlated with PET scan
  * d = number of subjects with no lesions detected by conventional scan or PET scan.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour, 2 hours post-injection)
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percent Agreement
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
Number analyzed (Participants) | 6 | 12 | 12
Percent Agreement
  PET(1hr): Positive percent agreement | 0.0 [NA to NA] — Not calculated, 0 participants with at least 1 positive lesion detected by conventional scan or at least 1 positive lesion detected by PET scan | 0.0 [NA to NA] — Not calculated, 0 participants with at least 1 positive lesion detected by conventional scan or at least 1 positive lesion detected by PET scan | 87.5 [47.35 to 99.68]
  PET(1hr): Negative percent agreement | 66.7 [22.28 to 95.67] | 25.0 [5.49 to 57.19] | 0.0 [0.00 to 60.24]
  PET(1hr): Overall percent agreement | 66.7 [22.28 to 95.67] | 25.0 [5.49 to 57.19] | 58.3 [27.67 to 84.83]
  PET(2hr): Positive percent agreement | 0.0 [NA to NA] — Not calculated, 0 participants with at least 1 positive lesion detected by conventional scan or at least 1 positive lesion detected by PET scan | 0.0 [NA to NA] — Not calculated, 0 participants with at least 1 positive lesion detected by conventional scan or at least 1 positive lesion detected by PET scan | 87.5 [47.35 to 99.68]
  PET(2hr): Negative percent agreement | 33.3 [4.33 to 77.72] | 25.0 [5.49 to 57.19] | 50.0 [6.76 to 93.24]
  PET(2hr): Overall percent agreement | 33.3 [4.33 to 77.72] | 5.49 [5.49 to 57.19] | 75.0 [42.81 to 94.51]

17. Secondary Outcome: Burden of Tumor Lesions Measured by 68Ga-PSMA-R2 PET (1hr) Scan Compared With Standard Imaging Modality, by Location (Overall)
Description: The differences of number of positive lesions, number of positive lesions detected by PET scan and/or conventional scan and the location of positive lesions were summarized with descriptive statistics.
Time Frame: 68Ga-PSMA-R2 PET imaging acquired at Day 1 (1 hour post-injection)
Population: Full Analysis Set (FAS)
Measure: Number; unit: Positive Lesion
Groups:
- Overall: All eligible participants received recommended dose of [68Ga]-PSMA-R2 of 3 Mega Becquerel (MBq)/Kg (+/- 10%) [but not more than 250 and not less than 150 MBq].
Arm/Group | Overall
Number analyzed (Participants) | 30
Positive Lesion
  PET (positive) | 22
  Conventional (postive) | 8
  Difference = PET(+) - Conventional(+) | 14
  PET(+) and detected by conventional scan | 7
  PET+/detected by CT:Bone,Cervical Spine | 1
  PET+/detected by CT:Bone,Lumbar Spine | 3
  PET+/detected by CT:Bone,Thoracic Spine | 3
  PET+/detected by CT:Pelvic Bone | 2
  PET+/detected by CT:Pelvis | 1
  PET+/detected by CT:Rib(s),L. | 1
  PET+/detected by CT:Rib(s),R. | 1
  PET(+) and not detected by conventional scan | 21
  PET+/undetected by CT:Abdominal Wall | 1
  PET+/undetected by CT:Bone,Lumbar Spine | 1
  PET+/undetected by CT:Bone,Other | 5
  PET+/undetected by CT:Bone,Thoracic Spine | 1
  PET+/undetected by CT:Lymph Node,Common Iliac | 9
  PET+/undetected by CT:Lymph Node,External | 1
  PET+/undetected by CT:Lymph Node,Inguinal,L. | 1
  PET+/undetected by CT:Lymph Node,Inguinal,R. | 1
  PET+/undetected by CT:Lymph Node,Para-Aortic | 6
  PET+/undetected by CT:Lymph Node,Retrocrural | 1
  PET+/undetected by CT:Lymph Node,Retroperitoneal | 2
  PET+/undetected by CT:Lymph Node,Supraclavicular,L | 1
  PET+/undetected by CT:Other,Extranodal | 3
  PET+/undetected by CT:Other,Nodal | 3
  PET+/undetected by CT:Pelvic Bone | 6
  PET+/undetected by CT:Rib(s),L. | 1
  PET+/undetected by CT:Rib(s),R. | 2
  PET+/undetected by CT:Urethra | 1
  Conventional (+) and not detected by PET scan | 7
  CT+/undetected by PET:Bone,Lumbar Spine | 2
  CT+/undetected by PET:Bone,Other | 2
  CT+/undetected by PET:Bone,Thoracic Spine | 5
  CT+/undetected by PET:Lymph Node,Pelvic | 1
  CT+/undetected by PET:Pelvic Bone | 6
  CT+/undetected by PET:Rib(s),L. | 2
  CT+/undetected by PET:Rib(s),R. | 1
  CT+/undetected by PET:Skull | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from informed consent signature through study completion, an average of 4 weeks.
Description: Any sign or symptom that occurs after written informed consent provided. For TEAE from first dosing (single administration, Day 1) up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the patient was lost to follow-up or withdrew consent.
Arm/Group | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) | Metastatic Prostate Cancer (mPCa) (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/6 | 4/12 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) (N=6) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) (N=12) | Metastatic Prostate Cancer (mPCa) (Phase II) (N=12)
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase I) (N=6) | Biochemically Recurrent Prostate Cancer (PCa-BR) (Phase II) (N=12) | Metastatic Prostate Cancer (mPCa) (Phase II) (N=12)
Fatigue (General disorders) | 0 | 2 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03490032/SAP_000.pdf
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03490032/Prot_001.pdf